CLINICAL TRIAL: NCT01589757
Title: The Effect of a Low GI Diet on Maternal and Neonatal Markers of Glycaemic Control and Postpartum Diabetes Risk SUBSTUDY The Effect of a Low GI Diet on Postpartum Markers of Oxidation in Breast Milk of Women With Gestational Hyperglycaemia
Brief Title: MAIN STUDY: Low Glycaemic Index (GI) Diet in the Management of GDM SUB-STUDY: The Breast Milk Sub-Study
Acronym: GIinGDM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Diabetes Association (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Foundation for Dietetic Research (CFDR) (Other)
Responsible Party: Principal Investigator, Thomas Wolever, Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UofTORE26937
Record Dates: First submitted 2012-04-19; First posted 2012-05-02 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Gestational Diabetes Mellitus
Keywords: "glycaemic index"; "glycemic index"; hyperglycaemia; hyperglycemia; pregnancy; "dietary intervention"; "education evaluation"; antioxidant; "Impaired Glucose Tolerance of Pregnancy"; "Gestational Diabetes Mellitus"; "Breast Milk"
MeSH Terms: conditions — Diabetes, Gestational; Hyperglycemia | interventions — Standard of Care; Glycemic Index

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Placebo Comparator): Standard care dietary advice to emphasize high fiber foods with a moderate to high GI
  Interventions: Other: Low GI diet
- Low GI Diet (Experimental): Low GI dietary advice in addition to standard care
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Standard Care — Standard dietary advice for women with GDM with special emphasis on use of high fiber or whole grain carbohydrate foods with a medium to high GI. What's on Your Plate? and 3-dimensional food models will be used to teach servings size and meal planning. This groups will be provided with food substitution lists (key-foods method) composed of medium to high GI foods.
  Other Names: medium to high Glycaemic Index
  Arms: Low GI Diet
Other: Low GI diet — Nutrition education according to standard care similar to the control group with supplementary GI-education. GI-education will be taught using the "Stop-Light-Method". This groups will be provided with food substitution lists (key-foods method) composed of low-GI carbohydrate-containing food. The GI-education tool(s) will build on standard care education where patients are taught which food groups contain carbohydrate.
  Other Names: glycemic index; glycaemic index; low glycemic carbohydrates; low glycaemic carbohydrates
  Arms: Standard Care

SUMMARY:
MAIN STUDY: Low glycaemic index (GI) diets are recommended by the Canadian Diabetes Association for treating type 1 and 2 diabetes mellitus (DM), but the role of GI in the management of gestational diabetes(GDM)is not yet clear. The main purpose of this study is to determine the effect of a low GI diet on blood sugar control in women with GDM. The effect of a low GI diet on maternal oxidative stress, pregnancy and delivery outcomes and markers of risk for diabetes after birth in both the mother and baby will also be assessed. SUB-STUDY: The main purpose of the sub-study is to determine if the breast milk (BM) of women with GDM consuming a low GI diet will have a higher antioxidant capacity than the BM of women receiving a medium-high GI diet (control/standard care). The effect of a low glycaemic index diet on maternal dietary intake of specific nutrient-antioxidants (i.e. vitamin C, E, and beta-carotene) (prenatal and postpartum) and concentration of vitamin C, E, and beta-carotene in participants' transitional and mature BM will also be assessed. The ORAC (Oxygen radical absorbance capacity) assay will be used to assess overall antioxidant capacity. The antioxidant capacity of BM in women with GDM will also be compared with that of women without GDM.

Hypotheses:

MAIN: The use of low-GI foods in the management of GDM reduces postprandial BG and oxidative stress; thereby reducing maternal and infant perinatal complications.

SUB-STUDY: Breast milk (BM) of women with GDM consuming a low GI diet will have higher BM antioxidant than women receiving the medium to high GI diet. BM of women with GDM will have lower antioxidant capacity than that of women without GDM.

DETAILED DESCRIPTION:
MAIN STUDY: Use of low GI education is currently accepted by the Canadian Diabetes Association in treatment of type 1 and 2 DM, but is not included in the clinical practice guidelines(CPG) for management of GDM. Data collected to date support use of low GI in treatment of GDM, but more data are needed to influence CPG. In this study the effect of a low GI diet on maternal and neonatal markers of glycaemic control and postpartum diabetes risk in mother and baby will be determined. This study will also assess the role that maternal oxidative stress may play in this relationship.

Hypothesis: The use of low-GI foods in the management of GDM reduces postprandial BG and oxidative stress; thereby reducing maternal and infant perinatal complications.

SUB-STUDY: Breast milk (BM) is accepted as the optimal source of nutrition for infants. A wealth of literature on BM composition exists. This work includes measurement of antioxidants in BM. Women diagnosed with gestational hyperglycaemia have decreased antioxidant capacity in comparison to normoglycaemic pregnant women. A direct relationship exists between postprandial glycaemic response and oxidative stress. Low GI carbohydrate is converted to blood glucose (BG) more slowly than medium to high GI carbohydrate

Hypotheses: Breast milk (BM) of women with GDM consuming a low GI diet will have higher BM antioxidant than women receiving the medium to high GI diet. BM of women with GDM will have lower anti-oxidant capacity than that of women without GDM.

ELIGIBILITY:
MAIN STUDY

Inclusion Criteria:

Women:

1. ≥ 18 years of age
2. diagnosed with gestational diabetes mellitus (GDM) or impaired glucose tolerance of pregnancy (IGTP) according to Canadian Diabetes Association (CDA) criteria
3. being followed within DIP (one of 4 sites)
4. willing and able to give informed consent
5. willing and able to comply with the study protocol

Exclusion Criteria:

Women:

1. with acute or chronic illness other than GDM or IGTP or use of drug (other than insulin) which may affect carbohydrate metabolism, gastrointestinal function or carbohydrate digestion (i.e. crohn's disease, HIV/AIDS, liver disease, kidney disease etc.).
2. known to have type 1 or type 2 DM prior to pregnancy
3. known multi-fetal pregnancy at enrolment
4. ≥ 33 weeks' gestation
5. prescribed oral anti-hyperglycaemic medication
6. insurmountable language barriers

SUB-STUDY control group (women without GDM) Same as for Main study except absence of GDM

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
MAIN STUDY: Percentage of postprandial self monitored blood glucose (SMBG) values within the target range | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the randomization to delivery. The endpoint is a single value for each participant - namely the percentage of all the postprandial SMBG values within the target range recommended by the Canadian Diabetes Association (5.0 to 6.6 mmol/L)
SUB-STUDY (n=75): Oxygen Radical Absorbance Capacity (ORAC) (Antioxidant Capacity) of transitional and mature breast milk. | 1 week and 8 weeks postpartum
  Breast milk samples (25 mL) will be collected 1 week and 8 weeks after birth from a complete breast milk collection. Measures will be compared between and within groups.

SECONDARY OUTCOMES:
MAIN STUDY: Infant birth weight | At delivery
  Weight of the baby at delivery in grams.
MAIN STUDY: Percentage of self-monitored fasting glucose values within the target range | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the start of the intervention to delivery. The endpoint is a single value for each participant - namely the percentage of all the fasting SMBG values within the target range recommended by the Canadian Diabetes Association (3.8 to 5.2 mmol/L)
MAIN STUDY: Glucose variability | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the randomization to delivery. This endpoint is the coefficient of variation of all the SMBG values obtained (CV = 100*SD/mean), where SD is standard deviation; a single value for each participant.
MAIN STUDY: Insulin prescription incidence | From randomization to delivery
  Proportion of women prescribed insulin during the intervention
MAIN STUDY: Mean fasting glucose | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the randomization to delivery. The endpoint is the mean of all fasting SMBG values obtained - a single value for each participant.
MAIN STUDY: Mean postprandial glucose | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the randomization to delivery. This endpoint is the mean of all postprandial SMBG values obtained; a single value for each participant.
MAIN STUDY: Mean post-breakfast glucose | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the randomization to delivery. This endpoint is the mean of all SMBG values 2 hours after breakfast; a single value in each participant.
MAIN STUDY: Mean post-lunch blood glucose | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the randomization to delivery. This endpoint is the mean of all SMBG values 2 hours after lunch; a single value in each participant.
MAIN STUDY: Mean post-dinner blood glucose | From randomization to delivery
  SMBG values are obtained 4 times daily (1 fasting and 3 postprandial) throughout the study from the randomization to delivery. This endpoint is the mean of all SMBG values 2 hours after dinner; a single value in each participant.
MAIN STUDY: Change in LDL oxidation at 4 weeks | Change from randomization in LDL oxidation at 4 weeks.
  Difference between LDL oxidation measured in fasting venous blood at randomization and 4 weeks.
MAIN STUDY: LDL oxidation 6-8 weeks after delivery | 6-8 weeks after delivery
  LDL oxidation measured in fasting venous blood 6-8 weeks after delivery.
MAIN STUDY: Change in Oxygen Radical Absorbance Capacity (ORAC) of plasma at 4 weeks | Change from randomization to 4 weeks
  Difference in Oxygen Radical Absorbance Capacity (ORAC) of plasma measured in venous serum at randomization and 4 weeks.
MAIN STUDY: Change in c-reactive protein (CRP) at 4 weeks | Change in CRP from randomization at 4 weeks
  Difference in c-reactive protein concentration in venous serum from baseline at 4 weeks.
MAIN STUDY: Post-partum CRP | 6-8 weeks after delivery
  Concentration of venous serum c-reactive protein 6-8 weeks after delivery.
MAIN STUDY: Post-partum fasting serum glucose | 6-8 weeks after delivery
  Venous fasting serum glucose 6-8 weeks after delivery
MAIN STUDY: Post-partum serum glucose concentration 2 hours after consumption of 75g oral glucose (2hrPC serum glucose). | 6-8 weeks after delivery
  Venous serum glucose concentration 2 hours after consumption of 75g oral glucose (oral glucose tolerance test).
MAIN STUDY: Incidence of post-partum impaired glucose tolerance | 6-8 weeks after delivery
  Proportion of women with venous serum glucose concentration 2 hours after a 75g oral glucose tolerance test between 7.8 and 11.0 mmol/L, inclusive.
MAIN STUDY: Incidence of post-partum diabetes mellitus | 6-8 weeks after delivery
  Proportion of women with diabetes 6-8 weeks after delivery. Diabetes is defined as fasting serum glucose greater than or equal to 7.0 mmol/L and/or serum glucose 2 hours after 75g oral glucose tolerance test greater than or equal to 11.1mmol/L.
MAIN STUDY: Maternal weight gain | From pre-pregnancy to delivery: up to 9 months
  Difference between reported pre-pregnancy body weight and last body weight measured before delivery.
MAIN STUDY: Rate of maternal weight gain | From randomization to delivery
  Difference between maternal body weight at randomization and last body weight measured before delivery divided by the number of weeks between the measurements.
MAIN STUDY: Change in infant weight | Change in infant body weight from birth to 6- 8 weeks
  Difference between infant birthweight and weight 6-8 weeks after delivery.
MAIN STUDY & SUB-STUDY (n=75): Maternal dietary intake | From randomization to 6- 8 weeks post-partum
  Dietary analysis will be conducted using software containing the Canadian Nutrient File, supplemented with data that used standardized GI testing methodology. Comparison will be made between and within groups.
SUB-STUDY (n=75): Concentration of vitamin C, E, and Beta-carotene in transitional breast milk | 1 week after delivery
  Concentration of vitamin C, vitamin E and beta-carotene in breast milk collected 1 week after delivery. Comparison will be made between and within study groups.
SUB-STUDY (n=75): Concentration of vitamin C, E, and Beta-carotene in mature breast milk | 6-8 weeks after delivery
  Concentration of vitamin C, vitamin E and beta-carotene in breast milk collected 6-8 weeks after delivery. Comparison will be made between and within study groups.
MAIN STUDY: Infant demographics | Delivery to 6-8 weeks postpartum
  Collection of infant demographics, such as gestational age at birth, sex, incidence and type of complications as noted in maternal or infant chart, mode of delivery, length of stay in hospital
MAIN STUDY: Change in infant body measurements from birth to 6-8 weeks post-partum | Change in infant body measurements from delivery to 6-8 weeks post-partum
  Weight, head circumference, and height/length
MAIN STUDY: Infant APGAR score at delivery | Delivery
  Infant APGAR score at delivery as recorded in maternal medical chart.
MAIN STUDY: Change in maternal blood pressure and resting pulse from randomization to 4 weeks | Change from randomization to 4 weeks.
  Difference between maternal blood pressure and resting pulse from randomization at4 weeks.
MAIN STUDY: Maternal blood pressure and resting pulse at 6-8 weeks post-partum | 6-8 weeks after delivery
  Maternal blood pressure and resting pulse at 6-8 weeks post-partum.
MAIN STUDY: Infant waist circumference at 6-8 weeks | 6-8 weeks after delivery
  Infant waist circumference at 6-8 weeks.
MAIN STUDY: Change in ultrasound measurements from randomization to delivery. | Change from randomization to delivery
  Difference between infant ultrasound measurements (Bi-parietal diameter, head circumference, abdominal circumference, and femur length) from baseline to delivery.
MAIN STUDY: Maternal height at baseline | Baseline
  Maternal height at baseline
MAIN STUDY: Maternal medical history | Baseline
  Maternal medical history
MAIN STUDY: Maternal medical complications from baseline to 6-8 weeks post-partum | Baseline to 6-8 weeks after delivery
  Incidence and type of maternal medical complications from baseline to 6-8 weeks post-partum
MAIN STUDY: Change in maternal weight from delivery at 6-8 weeks post-partum | Difference between delivery and 6-8 weeks post-partum
  Difference in maternal weight from delivery at 6-8 weeks postpartum.
MAIN STUDY: Maternal pre-natal demographic information | Baseline
  Maternal pre-natal demographic information (e.g. ethnicity, language used at home, household food preparation and purchasing, education obtained, employment status, treatment of diabetes, prior exposure to a registered dietitian, cigarette, recreational drug, and alcohol use before and during pregnancy, and physical activity) using a pre-tested, face-validated questionnaire.
MAIN STUDY: Maternal post-partum socio-demographic data related to infant feeding practices | 6-8 weeks after delivery
  Socio-demographic factors previously identified in the literature as affecting infant feeding practices; including access to breastfeeding education while in hospital.
MAIN STUDY: Length of time between delivery and maternal breast fullness | Time after delivery
  Length of time between delivery and maternal breast fullness.
MAIN STUDY: Change in conjugated dienes at 4 weeks | change from baseline to 4 weeks.
  Difference between conjugated dienes of plasma measured in venous serum at baseline and 4 weeks.
MAIN STUDY: Conjugated dienes post-partum | 6-8 weeks after delivery
  Conjugated dienes in fasting venous blood 6-8 weeks after delivery
MAIN STUDY: Oxygen Radical Absorbance Capacity (ORAC) of venous plasma post-partum | 6-8 weeks after delivery
  ORAC measured in fasting venous blood 6-8 weeks after delivery
MAIN STUDY: Change in full lipid profile at 4 weeks | Change in full lipid profile of plasma from baseline at 4 weeks
  Difference in full lipid profile of fasting venous blood at baseline and 4 weeks.
MAIN STUDY: Full lipid profile post-partum | 6-8 weeks after delivery
  Full lipid profile of fasting venous blood at 6-8 weeks post-partum
MAIN STUDY: Change in incidence and severity of symptoms from baseline to 6-8 weeks postpartum | Change from baseline to 6-8 weeks postpartum
  Difference in the incidence and severity of maternal symptoms present from baseline to 6-8 weeks postpartum using a standardised questionnaire.
MAIN STUDY: Infant feeding practices | 6-8 weeks after delivery
  Maternal infant feeding practices from delivery to 6-8 weeks postpartum
MAIN STUDY: Participant satisfaction of baseline education class | Baseline
  Participant reactions and opinions on baseline education class using a face-validated, pre-tested questionnaire.
MAIN STUDY: Change in participant knowledge of GI from baseline to 6-8 weeks after delivery | Change in GI knowledge from randomization to 6-8 weeks after delivery
  Difference in participant knowledge of GI from randomization pre-education class) to 6-8 weeks after delivery using a face-validated, pre-tested questionnaire.
MAIN STUDY: Participant knowledge of GI at baseline | Baseline
  Participant knowledge of GI at baseline (pre-education class)using a validated questionnaire.
MAIN STUDY: Change in participant opinion on availability and acceptability of study diet foods | Change in opinion from 2 weeks to 6-8 weeks after delivery
  Difference in participant opinion on availability and acceptability of study diet foods from 2 weeks to 6-8 weeks after delivery using a validated questionnaire.
MAIN STUDY: Difference in dietary GI between study groups. | From baseline to 6-8 weeks after delivery
  Difference in dietary GI between study groups from baseline to 6-8 weeks post delivery using a short-form semi-quantitative food frequency questionnaire (FFQ). The FFQ collects dietary intake data on the 3 months preceding administration. The FFQ has been standardised and evaluated for readability by nutrition professionals, clinicians and/or researchers with experience in surveying, and has been face-validated and pre-tested.
MAIN STUDY: Change in behaviour from baseline (pre-class) to 6-8 weeks after delivery. | Change in behaviour from baseline (pre-class) to 6-8 weeks after delivery
  Difference in behaviour within and between groups from baseline (pre-class) to 6-8 weeks after delivery using face-validated, pre-tested questionnaires, including a short-form semi-quantitative food frequency questionnaire (FFQ). The FFQ collects dietary intake data on the 3 months preceding administration. The FFQ has been standardised and evaluated for readability by nutrition professionals, clinicians and/or researchers with experience in surveying.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto/ St Michael's Hospital
Locations (4):
- Canada (4):
  - MAIN STUDY ONLY: St Joseph's Heathcare Hamilton, 50 Charlton Avenue East, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mt Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Background] Ceriello A. Acute hyperglycaemia and oxidative stress generation. Diabet Med. 1997 Aug;14 Suppl 3:S45-9. doi: 10.1002/(sici)1096-9136(199708)14:3+3.3.co;2-i. PMID 9272613
- [Background] Ceriello A. The emerging role of post-prandial hyperglycaemic spikes in the pathogenesis of diabetic complications. Diabet Med. 1998 Mar;15(3):188-93. doi: 10.1002/(SICI)1096-9136(199803)15:33.0.CO;2-V. No abstract available. PMID 9545118
- [Background] Huang D, Ou B, Prior RL. The chemistry behind antioxidant capacity assays. J Agric Food Chem. 2005 Mar 23;53(6):1841-56. doi: 10.1021/jf030723c. PMID 15769103
- [Background] Saenz AT, Elisia I, Innis SM, Friel JK, and Kitts DD. Use of ORAC to assess antioxidant capacity of human milk. Journal of Food Composition and Analysis 22:694-698, 2009
- [Background] Elisia I, Kitts DD. Quantification of hexanal as an index of lipid oxidation in human milk and association with antioxidant components. J Clin Biochem Nutr. 2011 Nov;49(3):147-52. doi: 10.3164/jcbn.10-142. Epub 2011 Sep 3. PMID 22128211
- [Background] Wolever, TMS. The Glycaemic Index: A Physiological Classification of Dietary Carbohydrate. Ontario, Canada: CABI, 2006.
- [Background] Grant SM, Wolever TMS. Perceived barriers to application of glycaemic index: valid concerns or lost in translation? Nutrients. 2011 Mar;3(3):330-340. doi: 10.3390/nu3030330. Epub 2011 Feb 28. PMID 22254100